CLINICAL TRIAL: NCT01627054
Title: A Phase II Study of AT7519M, a CDK Inhibitor, in Patients With Relapsed and/or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I193
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-03

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AT7519M (Experimental)
  Interventions: Drug: AT7519M

INTERVENTIONS:
Drug: AT7519M — Dose: 27 mg/m2, IV injection, 1 hour infusion Schedule: 27 mg/m2/day twice weekly x 2 weeks every 3 weeks (days 1, 4, 8 and 11)

SUMMARY:
The purpose of this study is to find out what effects a new drug AT7519M has on chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
This research is being done because AT7519M has been shown to shrink tumours in animals, has been studied in a few people and seems promising, but it is not clear if it can offer better results than standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previously documented CLL as defined by the 2008 International Workshop on Chronic Lymphocytic Leukemia guidelines [Hallek 2008(a)], that is recurrent or relapsed after previous therapy and that requires treatment.
* Patients must have a life expectancy of at least 12 weeks.
* Age ≥ 18 years.
* ECOG performance status of 0, 1 or 2
* Measurable disease criteria to assess response. Patients must have at least ONE of:

Absolute lymphocyte count ≥ 10 x 10^9/L OR At least one pathologically enlarged lymph node (≥ 2 x 2 cm) by CT scan

* Previous Therapy Patients must have received at least one, and may have received up to three prior systemic treatment regimens (single agent or combination therapy), there is no limit on number of prior regimens.

Systemic Therapy:

Patients must have received at least one prior systemic treatment regimen (single agent or combination therapy). There is no limit on number of prior regimens.

Patients must be ≥ 4 weeks since last dose of systemic therapy (including investigational). Exceptions to the 4-week interval since last treatment are possible if prior therapy is non-myelosuppressive or if any treatment-related myelosuppression has resolved.

Rationale:

Based on a review of recently published phase II trials of CDK inhibitors in relapsed and refractory CLL, there does not appear to be sufficient grounds to restrict the number of previous cycles of systemic chemotherapy. The IND193 investigators do not predict that this change will affect either the safety or efficacy outcomes of the study drug.

* Not permitted:
* Radioactive Monoclonal Antibody Therapy
* Prior treatment with AT7519M or another CDK inhibitor
* Previous allogeneic stem cell transplant (Note: autologous stem cell transplant is permitted)

Radiation:

Patients may have had radiation, provided a minimum of 21 days has elapsed prior to enrollment. (Exceptions may be made however, for low dose, palliative radiotherapy Patients must have recovered from any acute toxic effects from radiation prior to registration.

Surgery:

Previous surgery is permitted provided that wound healing has occurred and at least 14 days have elapsed if surgery was major.

* Laboratory Requirements: (must be done within 7 days prior to registration) Hematology = Absolute neutrophils (ANC) ≥ 1.0 x 10^9/L Platelets = ≥ 75 x 10^9/L (exception: if ITP secondary to CLL, allow 50 x 10^9/L) Chemistry = Creatinine clearance* ≥ 50 mL/min Creatine Phosphokinase = (CK or CPK) ≤ UNL Bilirubin = ≤ UNL AST and ALT = ≤ 2.5 x UNL Potassium, Calcium, Magnesium Within normal limits
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is provided as a separate attachment. A copy of the initial REB approval and approved consent form must be sent to the central office. The patient must sign the consent form prior to registration. Please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient registration.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, other in situ cancers or other invasive malignancies curatively treated with no evidence of disease for ≥ 5 years.
* Patients with known CNS involvement by CLL. Tests to investigate CNS involvement are required only if clinically indicated (i.e. disease suspected on basis of symptoms or other findings).
* Patients with clinically suspected or proven progression to high grade lymphoma (Richter's transformation) or myelodysplasia.
* Patients with known hypersensitivity to the study drug or its components.
* The following are exclusions for enrolment on the study:

  1. Pregnant or lactating women. (N.B.: All women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to registration).
  2. Men and women of childbearing potential who do not agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of the study participation. (Should a woman become pregnant or suspect she is pregnant, or should a man father a child, while participating in this study, she/he should inform the treating physician immediately.)
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including, but not limited to:

  1. history of significant neurologic or psychiatric disorder (e.g. uncontrolled psychotic disorders) which would impair the ability to obtain consent or limit compliance with study requirements;
  2. active uncontrolled or serious infection (viral, bacterial or fungal);
  3. pulmonary disease requiring oxygen;
  4. known HIV infection or other immune deficiency disorders (except for CLL);
  5. other medical conditions that might be aggravated by study treatment
* Patients with pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction as follows:

  1. Significant cardiac event (including heart failure or ischemia) within 3 months of entry or any cardiac disease that, in the opinion of the investigator, increases risk for ventricular arrhythmia
  2. Any family or personal history of ventricular arrhythmia, which was symptomatic or required treatment (CTC grade 3). This includes: multifocal PVCs, bigeminy, trigeminy, ventricular tachycardia)
  3. Uncontrolled hypertension (systolic blood pressure of 150 mmHg or higher or diastolic blood pressure of 95 mmHg or higher)
  4. A previous history of drug induced QTc prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant ECG abnormalities
  5. Congenital long QT syndrome
  6. QT and QTc, unmeasurable or > 460 msec on screening ECG
  7. Left ventricular ejection fraction (LVEF) of less than the institution's lower limit of normal (LLN) measured by MUGA or echocardiogram
* Patients who are currently receiving treatment with agents with a known risk of Torsades de Pointes. (see http://torsades.org [list #1]). However, patients may be enrolled on study if treatment with such agents is stopped ≥ 7 days prior to first dose of AT7519M.
* Patients with pre-existing peripheral neuropathy (sensory and/or pain) > grade 2.
* Patients with uncontrolled auto-immune hemolytic anemia (AIHA) and/or auto-immune thrombocytopenia (ITP) who require active treatment.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2014-03-21 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 24 months
  Efficacy (as assessed by objective response rate) of AT7519M when given as a 1 hour intravenous infusion twice weekly for two out of three weeks in patients with relapsed and/or refractory chronic lymphocytic leukemia.

SECONDARY OUTCOMES:
Toxicity severity | 24 months
Time to progression | 24 months
Response duration | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Seftel, Study Chair — Cancer Care Manitoba, Winnipeg Manitoba Canada
Locations (3):
- Canada (3):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seftel MD, Kuruvilla J, Kouroukis T, Banerji V, Fraser G, Crump M, Kumar R, Chalchal HI, Salim M, Laister RC, Crocker S, Gibson SB, Toguchi M, Lyons JF, Xu H, Powers J, Sederias J, Seymour L, Hay AE. The CDK inhibitor AT7519M in patients with relapsed or refractory chronic lymphocytic leukemia (CLL) and mantle cell lymphoma. A Phase II study of the Canadian Cancer Trials Group. Leuk Lymphoma. 2017 Jun;58(6):1358-1365. doi: 10.1080/10428194.2016.1239259. Epub 2016 Oct 17. PMID 27750483